CLINICAL TRIAL: NCT01967602
Title: Biomarker of Lung Injury in ARDS Patients Receiving ECMO Support
Acronym: ARDS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201103056RB
Record Dates: First submitted 2013-10-18; First posted 2013-10-23 (Estimated); Last update posted 2013-10-23 (Estimated); Status verified 2013-10

CONDITIONS: ARDS; Multi-organ Failure
Keywords: Acute respiratory distress syndrome (ARDS); Extracorporeal membrane oxygenation (ECMO); biomarker
MeSH Terms: conditions — Multiple Organ Failure; Respiratory Distress Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Plasma, Cell, BALF, Urine
Oversight: Data Monitoring Committee: No

SUMMARY:
The goal of this project is to find a marker expression that the investigators can use to trace symptom progression and develop a more efficient therapy to enhance ARDS patient survival rate and better post-ICU life quality.

DETAILED DESCRIPTION:
The investigators will first identify acute respiratory distress syndrome (ARDS) patients receiving ECMO support in ICU at National Taiwan University Hospital, and then collect blood, urine and bronchioalveolar lavage fluid (BALF) samples at different time points: before setting up ECMO, 2, 6, 12, 24, 72 hours,5 and 14 days after ECMO installment, time to wean ECMO and the day removing ECMO and leaving ICU. From the samples, the free radicals, cytokines (IL-1, IL-6, IL-8, IL-18,tumor necrosis factor-α, transforming growth factor-β), and inflammasome- related markers, immune cell responses and other biochemical markers would be measured. The novel biomarkers to predict the outcome of the patient will be identified.

ELIGIBILITY:
Inclusion Criteria:

1. >18 years old
2. ARDS, needing ECMO support

Exclusion Criteria:

1. pre-existing sepsis
2. pre-existing chronic renal failure (dialysis dependent), liver failure other diseases precluding chance of survival.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who are admitted to National Taiwan University Hospital for acute respiratory distress syndrome needing ECMO placement.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2011-10; Primary Completion 2015-04 (Estimated); Study Completion 2015-04 (Estimated)

PRIMARY OUTCOMES:
Mortality or multi-organ failure | 7 days
  Patients who survived for more than 7 days after ECMO treatment were defined as survival, and non-survival patients were defined as expired or multiple organ failure incompatible with life within 7 days after ECMO installation.

CONTACTS AND LOCATIONS:
Overall Officials: Shuenn-Wen Kuo, MD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan